CLINICAL TRIAL: NCT05972954
Title: A Phase 2a Safety, Tolerability, and Pharmacodynamic Study of OMT-28 in PMD Patients With Myopathy and/or Cardiomyopathy and Inflammation (PMD-OPTION)
Brief Title: OMT-28 in Patients With Primary Mitochondrial Disease (PMD) (PMD-OPTION)
Acronym: PMD-OPTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omeicos Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMT28-C0203
Record Dates: First submitted 2023-06-27; First posted 2023-08-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Primary Mitochondrial Disease
Keywords: Myopathy; Cardiomyopathy; Mitochondrial encephalopathy, lactic acidosis and stroke-like episodes (MELAS) syndrome; Myoclonic epilepsy with ragged red fibers (MERRF); Maternally inherited diabetes and deafness (MIDD) syndrome; GDF-15
MeSH Terms: conditions — Muscular Diseases; Cardiomyopathies; Mitochondrial encephalopathy; Acidosis, Lactic; MELAS Syndrome; Syndrome; MERRF Syndrome; Deafness; Noninsulin-dependent diabetes mellitus with deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with OMT-28 (Experimental): 24mg OMT-28, oral capsule, for 12 weeks
  Interventions: Drug: OMT-28

INTERVENTIONS:
Drug: OMT-28 — once daily

SUMMARY:
The goal of this clinical trial is to learn about the treatment effects of the investigational new drug OMT-28 in patients with Primary Mitochondrial Disease.

The main question[s] it aims to answer are:

* Is OMT-28 safe and well tolerated in this patient population?
* Does OMT-28 reduce Growth Differentiation Factor 15 (GDF-15) and other relevant blood markers of mitochondrial dysfunction and inflammation?
* Does OMT-28 improve symptoms of the disease, e.g. fatigue or exercise intolerance?

Participants will be asked to participate in 6 study visits at an experienced clinical center, including physical examinations and exercise tests, and take the study medication regularly once per day according to the protocol.

Researchers will compare for every participant the results after 3 months and 6 months of treatment with a preceding 3 month period of standard care treatment to investigate the effects of OMT-28 on clinical parameters and a number of blood parameters.

DETAILED DESCRIPTION:
This is an open label, single-arm, multiple-phase and multicenter Phase 2a study to evaluate the efficacy, safety, and pharmacokinetics of a single OMT-28 dose (24 mg given once daily) in patients with Primary Mitochondrial Disease and clinical manifestation of myopathy and/or cardiomyopathy.

Patients are eligible if they have

* Primary Mitochondrial Disease with a documented mitochondrial transfer ribonucleic acid (tRNA) point mutation, including m3243A>G, m8344A>G, or single mitochondrial DNA (mtDNA) deletions,
* a clinically relevant myopathy and/or cardiomyopathy confirmed following standard guidelines,
* a blood plasma GDF-15 concentration > 1200 ng/L and < 10.000 ng/L at screening

Participation in the study is divided into 3 parts:

* Screening and baseline: 12 weeks
* Treatment: 24 weeks
* Safety follow-up: 4 weeks

Total duration: 40 weeks

Safety will be monitored throughout the study. Blood samples for safety, pharmacodynamics and pharmacokinetics will be collected at every of the 6 study visits. Exercise tests (6/12-minutes walking test, 5xSST), transthoracic echocardiography, patient reported outcomes (e.g. Fatigue Severity Scale and Patients' Global Impression of Change (PGIC) scale) will be assessed at prespecified visits. Patients will be provided with a diary to record timing of drug administration and clinical symptoms while not on site. Diaries will be reviewed and checked for compliance at each non-resident visit to the clinical site.

ELIGIBILITY:
Inclusion Criteria:

1. Documented mutation resulting in mitochondrial disease: mitochondrial tRNA point mutations, including m3243A>G, m8344A>G, and single mtDNA deletions
2. Diagnosis of Cardiomyopathy defined as LV hypertrophy and/or LVEF<50% and/or late gadolinium enhancement on cardiac MRI and/or Myopathy as defined by the International Workshop: Outcome measures and clinical trial readiness in primary mitochondrial myopathies in children and adult (Mancuso et al. 2017[8])
3. GDF-15 between 1,200 ng/L and 10,000 ng/L at screening
4. Ability to perform the exercise tests

6. Willing and able to provide a signed Informed Consent, as well as written documentation in accordance with country and local privacy requirements, e.g., written data protection consent 7. Able and willing to comply with the requirements of this study protocol 8. Both female patients, as well as, female partners of male patients who are of child-bearing potential must be willing to not become pregnant for the complete duration of the study (30 days after the last dose of study medication).

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
3. Subjects with a history of cancer in the last 5 years
4. Hypertension defined as systolic BP >160 mmHg or diastolic BP >100 mmHg at screening
5. Uncontrolled Diabetes mellitus according to investigator's assessment
6. Stroke-like episodes or seizures occurred within last 6 months
7. Motoric abnormalities other than related to the mitochondrial disease interfering with the outcome parameters
8. History or evidence of active tuberculosis (TB) infection, any co-disease with inflammatory condition (e.g., Inflammatory Bowel Disease (IBD) etc.)
9. Patients with a positive hepatitis panel and/or positive immunodeficiency virus test at screening
10. Regular use of steroid, non-steroidal anti-inflammatory drug (NSAID), or colchicine within 30 days before screening
11. Chronic use of Metformin
12. Use of fish oil / omega-3 fatty acid supplements within two weeks before screening
13. Drinking more than 9 standard cups of alcohol per week and/or more than 3 standard cups of alcohol per occasion
14. Positive drug and alcohol screen (including opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines)
15. Any significant hepatic disease
16. Receiving any investigational therapy or any approved therapy for investigational use within 30 days or 5 half-lives prior to screening (whichever is longer)
17. Received any vaccines (including the booster vaccination for COVID-19) within two weeks prior to Visit 1
18. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study unless they agree to use adequate contraception as described in Appendix 11.4
19. Males (including sterilized subjects) and whose female partners have child-bearing potential, must agree to use male contraception (condoms) during the period from the time of signing the informed consent form (ICF) through 30 days after the last dose of study drug. They must agree to immediately inform the investigator if his partner becomes pregnant during the study
20. Subjects who have previously been exposed to OMT-28, whether responder or non-responder.
21. Any use of statins (HMG-CoA reductase inhibitors)
22. Use of quinine, tacrolimus, mycophenolate mofetil, ciclosporin, serotine receptor-type 1 agonist, penicillin G, penicillamine (d-penicillamine), nicotinic acid (niacin), colchicine, isotretinoin, and amiodarone, peroxisome proliferator-activated receptor (PPAR) activators, AMP-activated protein kinase (AMPK) activators, sirtuin activators, steroids, cyclooxygenase inhibitors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Responder rate | 12 weeks treatment vs. 12 weeks baseline
  Number of patients (responder rate) with a between phase difference in GDF-15 of at least 20% decrease
Number of Treatment Emergent Adverse Events (TEAE) | up to 28 weeks
  Compare the number of TEAEs during and between evaluation phases

SECONDARY OUTCOMES:
Responder rate | 24 weeks treatment vs. 12 weeks baseline
  Number of patients (responder rate) with a between phase difference in GDF-15 of at least 20%
Change in plasma concentration of GDF-15 [ng/L] | 12 weeks treatment vs. 12 weeks baseline
  GDF-15 plasma concentration during evaluation phases, change in GDF-15 concentration during evaluations phases and comparison of GDF-15 concentration between evaluation phases
Pharmacokinetics: Ctrough [ng/ml] | weeks 12, 16, 24 and 28
  Trough plasma concentrations (Ctrough) of OMT-28
Pharmacokinetics: Cmax [ng/ml] | week 12 and week 24
  Plasma concentration of OMT-28 approximately at Cmax and one further timepoint after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fischer, MD, Study Director — Omeicos Therapeutics GmbH
Locations (9):
- Germany (3):
  - Universitätsklinikum Bonn, Sektion Neuromuskuläre Erkrankungen, Klinik und Poliklinik für Neurologie, Venusberg-Campus 1, Gebäude 80, NPP, Bonn
  - Medizinisch Fakultät der Martin-Luther-Universität Halle-Wittenberg Universitätsklinik und Poliklinik für Neurologie Universitätsklinikum , Ernst-Grube-Str. 40, Halle
  - Friedrich-Baur-Institut an der Neurologischen Klinik und Poliklinik, Klinikum der Universität München, Ludwig-Maximilians-Universität (LMU Klinikum), Ziemssenstr. 1a, Munich
- Italy (5):
  - IRCCS Institute of Neurological Science of Bologna, University of Bologna, Department of Biomedical and Neuromotor Science (DIBINEM), Ospedale Bellaria Via Altura, 3, Bologna
  - U.O.C. di Neurologia e Malattie Neuromuscolari, Messina
  - IRCCS Istituto Neurologico Carlo Besta, SC Servizio Di Medicina Di Laboratorio - Genetica Medica E Neurogenetica, Via Celoria 11, Milan
  - Azienda Ospedaliero Universitaria Pisana, P.O. Santa Chiara, U.O. Neurologia, Edificio 13, Via Roma 67, Pisa
  - UOC di neurofisiopatologia, Roma
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands